CLINICAL TRIAL: NCT07274852
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of Lutetium [177Lu]-BL-ARC001 Injection in Patients With Locally Advanced or Metastatic Lung Cancer, Breast Cancer, Head and Neck Squamous Cell Carcinoma and Other Solid Tumors
Brief Title: A Study of Lutetium [177Lu]-BL-ARC001 in Patients With Locally Advanced or Metastatic Lung Cancer, Breast Cancer, Head and Neck Squamous Cell Carcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-BL-ARC001-101
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Breast Cancer; Head and Neck Squamous Cell Carcinoma; Solid Tumors
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Lutetium; Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lutetium [177Lu] BL-ARC001 (Experimental): Participants receive Lutetium [177Lu] BL-ARC001 for the first cycle (6 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Lutetium [177Lu] BL-ARC001

INTERVENTIONS:
Drug: Lutetium [177Lu] BL-ARC001 — Administration by intravenous infusion for a cycle of 6 weeks.

SUMMARY:
This study is an open, multicenter, dose-escalation and cohort-expansion non-randomized phase I clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of Lutetium [177Lu] BL-ARC001 in patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study is divided into two stages: the dose-escalation phase (Phase Ia) and the cohort-expansion phase (Phase Ib).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years (Phase Ia); ≥18 years (Phase Ib);
4. Expected survival time ≥3 months;
5. Histologically or cytologically confirmed locally advanced or metastatic solid tumors that have failed standard treatment;
6. Agreement to provide archived tumor tissue specimens or fresh tissue samples from primary or metastatic lesions within the past 3 years;
7. Must have at least one measurable lesion as defined by RECIST v1.1;
8. ECOG performance status score of 0 or 1;
9. Toxicity from prior antitumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. Organ function levels must meet the requirements;
12. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
13. Urine protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women with childbearing potential, a serum pregnancy test must be performed within 7 days before starting treatment, and the result must be negative. Patients must not be breastfeeding; all enrolled patients (regardless of gender) should adopt adequate barrier contraception throughout the treatment cycle and for 6 months after treatment ends.

Exclusion Criteria:

1. Use of chemotherapy, biological therapy, or immunotherapy within 4 weeks or 5 half-lives prior to the first dose;
2. History of severe heart disease;
3. Prolonged QT interval, complete left bundle branch block, or third-degree atrioventricular block;
4. Active autoimmune or inflammatory diseases;
5. Diagnosis of other malignancies within 5 years prior to the first dose;
6. Hypertension poorly controlled by two antihypertensive medications;
7. History of interstitial lung disease (ILD) requiring hormonal therapy, current ILD, or ≥ Grade 2 radiation pneumonitis;
8. Symptoms of active central nervous system metastasis;
9. History of allergy to recombinant humanized antibodies or human-mouse chimeric antibodies, or allergy to any excipient component of 177Lu-BL-ARC001;
10. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
11. Cumulative dose of anthracyclines >360 mg/m² during prior (neo)adjuvant anthracycline therapy;
12. Positive human immunodeficiency virus (HIV) antibody, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
13. Active infection requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
14. Participation in another clinical trial within 4 weeks prior to the first dose;
15. Pregnant or lactating women;
16. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 42 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 42 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of Lutetium [177Lu] BL-ARC001.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of Lutetium [177Lu] BL-ARC001. The type, frequency and severity of TEAE will be evaluated during the treatment of Lutetium [177Lu] BL-ARC001.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of Lutetium [177Lu] BL-ARC001 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of Lutetium [177Lu] BL-ARC001 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of Lutetium [177Lu] BL-ARC001 will be investigated.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of Lutetium [177Lu] BL-ARC001 per unit of time will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of Lutetium [177Lu] BL-ARC001 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-Lutetium [177Lu] BL-ARC001 antibody (ADA) will be investigated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China